CLINICAL TRIAL: NCT02320253
Title: REAL HEALTH-Diabetes: Reach Ahead for Lifestyle and Health-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Linda M. Delahanty, Chief Dietitian at Massachusetts General Hospital Diabetes Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P002074; 1R18DK102737-01A1 (NIH)
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Diabetes; Obesity; Primary Care; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical Nutrition Therapy (MNT) (Active Comparator): Participants in this arm will meet with a dietitian at their respective Health Center, not with a study dietitian. The participant and dietitian will decide how frequently to meet and create an individualized treatment plan. The participant's health insurance will be billed for these dietitian visit(s) and the participant is responsible for any copay(s) or deductible(s) associated with the visit(s).
  Interventions: Behavioral: Medical Nutrition Therapy (MNT)
- In Person Group (IP) (Experimental): Participants enrolled to the IP arm will meet weekly for 14 weeks, biweekly for 10 weeks, and then monthly for the next 18 months. Each session will be led by a study dietitian that has been assigned to that specific health center and will last 1.5 hours. Participants will be allowed to have one-on-one sessions with their dietitian throughout the first two years, twice in the first year and three times in the second year.
  Interventions: Behavioral: In Person Group (IP)
- Telephone Conference Call Group (TCC) (Experimental): Participants enrolled in the TCC arm will meet weekly for 14 weeks, biweekly for 10 weeks, and then monthly for the next 18 months. Each session will be led, over-the-phone, by a study dietitian that has been assigned to that specific health center and will last 1.5 hours. Participants will be allowed to have one-on-one sessions with their dietitian throughout the first two years, twice in the first year and three times in the second year.
  Interventions: Behavioral: Telephone Conference Call Group (TCC)

INTERVENTIONS:
Behavioral: In Person Group (IP) — The goals of the diabetes lifestyle intervention program are weight loss of 5-10% of initial body weight and increased activity levels to 175 minutes/week of moderate intensity physical activity. Dietitians will deliver the adapted Look AHEAD lifestyle intervention via in-person groups combined with 2-3 individual sessions per year. The program curriculum focuses on nutrition, activity, and behavioral topics and incorporates the use of meal replacements for the first 4-16 weeks to enhance weight loss success.
  Arms: In Person Group (IP)
Behavioral: Telephone Conference Call Group (TCC) — The goals of the diabetes lifestyle intervention program are weight loss of 5-10% of initial body weight and increased activity levels to 175 minutes/week of moderate intensity physical activity. Dietitians will deliver the adapted Look AHEAD lifestyle intervention via telephone conference call groups combined with 2-3 individual sessions per year. The program curriculum focuses on nutrition, activity, and behavioral topics and incorporates the use of meal replacements for the first 4-16 weeks to enhance weight loss success. Dietitians will deliver the adapted Look AHEAD lifestyle intervention.
  Arms: Telephone Conference Call Group (TCC)
Behavioral: Medical Nutrition Therapy (MNT) — Participants are referred to meet with a registered dietitian for individual medical nutrition therapy sessions up to 3-4 times per year.
  Arms: Medical Nutrition Therapy (MNT)

SUMMARY:
The goal of this project is to translate the Look AHEAD intensive lifestyle intervention for type 2 diabetes and obesity into usual care at community health centers, comparing an in-person group program (IP), a telephone conference call (TCC) group program, and referral to medical nutrition therapy (MNT), the current standard of care.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three arms: MNT, IP, or TCC. Participants will be enrolled in the study for a total of three years. During those three years, participants will have 5 research visits, at baseline, where randomization occurs, 6 months, 12 months, 24 months, and 36 months. At each research visit, participants will have a lipid panel and HbA1c sample drawn, their blood pressure, weight, and height, baseline only, taken. Participants will also answer questionnaires that will address health behaviors, self-efficacy, measures of self-determination, depression, literacy and numeracy, food insecurity, health-related quality-of-life and patient satisfaction with quality of care.

For the group-based interventions, dietitians will deliver the adapted Look AHEAD lifestyle intervention. The first 14 sessions will be delivered weekly and the next 5 sessions biweekly. In the subsequent 18 months, group sessions will be delivered monthly from 6-24 months. In addition, participants will be offered up to 5 individual MNT sessions over the 2 year intervention period. At these individual visits, dietitians will address diabetes-related issues and discuss tailored goals and behaviors, based on the Look AHEAD model. Dietitians will provide ongoing feedback to participants' own PCPs about patient progress toward goals and will encourage PCPs to reinforce weight loss strategies with their patients. Each group will contain up to 12 participants with type 2 diabetes and will last 1-1.5 hours. The program curriculum focuses on nutrition, activity, and behavioral topics and incorporates the use of meal replacements for the first 4-16 weeks to enhance weight loss success.

In addition to the teaching component, participants who are taking insulin or medications that can cause hypoglycemia will self-monitor blood glucose levels at least 2 times per day and submit self-monitoring records for review each week, either by delivering them at the in-person sessions or by mailing, faxing, or emailing them to the study team. Patients on oral hypoglycemics who are not adjusting medications based on blood sugar will be instructed to do targeted monitoring to determine the effects of exercise and meals on blood glucose. The study provider at each health center will review BG records and make any needed adjustments to insulin or medication doses according to an algorithm to maintain glycemic control and prevent hypoglycemia as participants lose weight.

A trained member of the study staff will provide MNT referral participants with an educational handout emphasizing that modest weight loss (5 - 10%) via caloric restriction and gradual adoption of moderate increases in daily physical activity (equivalent to brisk walking for 30 minutes daily) is safe and effective in managing diabetes and schedule them for an appointment with a dietitian from Nutrition Services for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Age 18 years or older
* Overweight or obese (BMI >25 kg/m2)
* HbA1c level 6.5<11.5%
* Systolic blood pressure (SBP) <160 mmHg, diastolic blood pressure (DBP) <100 mmHg
* Willing to lose 5-7% of body weight
* Willing to increase activity to at least 175 minutes/week
* Willing to commit to random assignment to either attend and participate in the lifestyle change program in person or on the telephone or be referred to Nutrition Services for medical nutrition therapy
* Stable health, with no severe comorbidities that might interfere with their ability to participate in a group intervention that includes increasing activity or decreasing calories, such as severe psychiatric illness or significant heart disease
* Ability to understand and communicate effectively in English or Spanish
* Willing to self-monitor blood glucose
* Willing to keep a food, exercise, and blood glucose diary
* Have a primary care physician at MGH Chelsea, Charlestown, or Revere Health Centers, or be willing to attend sessions, in-person or by phone, and have medications adjusted by a provider based at one of those health centers with communication to the referring primary care provider

Exclusion Criteria:

* Weight greater than 350 pounds
* Pregnant or planning pregnancy in the next year
* Currently seeing a dietitian (regular scheduled follow up appointments) or participating in a weight loss program and unwilling to stop
* Weight change of more than 3% of weight in the previous month.
* Currently enrolled in another diabetes intervention study
* Lack of availability of telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-11; Primary Completion 2020-09 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Delahanty, MS RD, Principal Investigator — Massachusetts General Hospital; Deborah J Wexler, MSc MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Charlestown HealthCare Center, Charlestown, Massachusetts
  - Chelsea HealthCare Center, Chelsea, Massachusetts
  - Revere HealthCare Center, Revere, Massachusetts

REFERENCES:
- [Background] Delahanty LM, Chang Y, Levy DE, Porneala B, Dushkin A, Bissett L, Goldman V, Perrotta J, Rodriguez AR, Chase B, LaRocca R, Wheeler A, Wexler DJ. Design and participant characteristics of a primary care adaptation of the Look AHEAD Lifestyle Intervention for weight loss in type 2 diabetes: The REAL HEALTH-diabetes study. Contemp Clin Trials. 2018 Aug;71:9-17. doi: 10.1016/j.cct.2018.05.018. Epub 2018 May 25. PMID 29803816
- [Derived] Vakharia JD, Thaweethai T, Licht P, Wexler DJ, Delahanty LM. Psychological and Behavioral Predictors of Weight Loss in the Reach Ahead for Lifestyle and Health-Diabetes Lifestyle Intervention Cohort. J Acad Nutr Diet. 2023 Jul;123(7):1033-1043.e1. doi: 10.1016/j.jand.2023.02.018. Epub 2023 Mar 5. PMID 36871848
- [Derived] Wexler DJ, Chang Y, Levy DE, Porneala B, McCarthy J, Rodriguez Romero A, Goldman V, Copeland PM, Steppel-Reznik J, Delahanty LM. Results of a 2-year lifestyle intervention for type 2 diabetes: the Reach Ahead for Lifestyle and Health-Diabetes randomized controlled trial. Obesity (Silver Spring). 2022 Oct;30(10):1938-1950. doi: 10.1002/oby.23508. Epub 2022 Aug 31. PMID 36046939
- [Derived] Berkowitz SA, Chang Y, Porneala B, Cromer SJ, Wexler DJ, Delahanty LM. Does the effect of lifestyle intervention for individuals with diabetes vary by food insecurity status? A preplanned subgroup analysis of the REAL HEALTH randomized clinical trial. BMJ Open Diabetes Res Care. 2020 Sep;8(1):e001514. doi: 10.1136/bmjdrc-2020-001514. PMID 32978121
- [Derived] Delahanty LM, Levy DE, Chang Y, Porneala BC, Goldman V, McCarthy J, Bissett L, Rodriguez AR, Chase B, LaRocca R, Wheeler A, Wexler DJ. Effectiveness of Lifestyle Intervention for Type 2 Diabetes in Primary Care: the REAL HEALTH-Diabetes Randomized Clinical Trial. J Gen Intern Med. 2020 Sep;35(9):2637-2646. doi: 10.1007/s11606-019-05629-9. Epub 2020 Jan 21. PMID 31965526
- [Derived] Goldman V, Dushkin A, Wexler DJ, Chang Y, Porneala B, Bissett L, McCarthy J, Rodriguez A, Chase B, LaRocca R, Wheeler A, Delahanty LM. Effective recruitment for practice-based research: Lessons from the REAL HEALTH-Diabetes Study. Contemp Clin Trials Commun. 2019 May 1;15:100374. doi: 10.1016/j.conctc.2019.100374. eCollection 2019 Sep. PMID 31193095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual enrollment 211
Period: Overall Study
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Started | 69 | 70 | 72
Completed | 63 | 68 | 70
Not Completed | 6 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Three participants from the MNT arm withdrew consent and were not analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC) | Total
Number analyzed (Participants) | 66 | 70 | 72 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.7) | 61.3 (10.3) | 62.4 (9.8) | 61.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 41 | 115
  Male | 29 | 33 | 31 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 7 | 28
  Not Hispanic or Latino | 55 | 60 | 65 | 180
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 2 | 9
  White | 47 | 55 | 58 | 160
  More than one race | 12 | 10 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Boston, MA, USA and surrounding communities
  participants
    United States | 66 | 70 | 72 | 208
Weight [Mean (Standard Deviation); unit: kg] — Weight is measured in kilograms.
  kg | 99.7 (21.4) | 98.8 (17.0) | 96.1 (18.2) | 98.7 (18.9)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 7.8 (1.2) | 7.8 (1.2) | 7.6 (1.1) | 7.7 (1.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure is measured in mmHg
  mmHg | 125 (16) | 126 (14) | 124 (10) | 125 (14)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 146 (99) | 196 (290) | 152 (94) | 165 (186)
Diet self efficacy scale [Mean (Standard Deviation); unit: units on a scale] — The Diet Self-Efficacy Scale ranges from 1-5 with higher scores denoting greater self confidence in measuring diet. Hickey ML, Owen SV, Froman RD. Instrument development: cardiac diet and exercise self-efficacy. Nursing research. 1992;41(6):347-51.
  units on a scale | 3.7 (0.6) | 3.6 (0.7) | 3.8 (0.7) | 3.7 (0.7)
Fat-related diet behavior [Mean (Standard Deviation); unit: units on a scale] — Fat-related diet behavior is graded from 1-5, in which lower scores indicate lower fat dietary habits. Kristal AR, Shattuck AL, Henry HJ. Patterns of dietary behavior associated with selecting diets low in fat: reliability and validity of a behavioral approach to dietary assessment. J Am Diet Assoc. 1990;90(2):214-20.
  units on a scale | 2.7 (0.6) | 2.7 (0.5) | 2.8 (0.6) | 2.7 (0.6)
Dietary restraint [Mean (Standard Deviation); unit: units on a scale] — Dietary restraint was measured by the Dutch Eating Behavior Questionnaire with higher scores (1-5) denoting greater self-regulation of dietary behaviors and positive values denoting improved dietary restraint. Van Strien T, Frijters JER, Defares PB. The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International Journal of Eating Disorders. 1986;5(2):295-315.
  units on a scale | 2.8 (0.6) | 2.9 (0.6) | 2.8 (0.8) | 2.8 (0.7)
Diabetes Distress [Mean (Standard Deviation); unit: score] — Diabetes distress was measured with the Problem Areas in Diabetes Scale, in which higher scores indicate greater emotional distress on a scale of 1 to 100, with a score of 40 marking the threshold for severe emotional distress. Negative values indicate reduction in diabetes-related distress. Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997;20(5):760-766
  score | 36.9 (23.1) | 39.3 (19.5) | 40.3 (23.3) | 38.9 (22.0)
Mood [Mean (Standard Deviation); unit: units on a scale] — The PHQ-8 measures depressed mood, with higher scores representing a higher degree of depressed mood and negative values indicating improvement. Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009;114(1-3):163-173.
  units on a scale | 5.3 (5.4) | 4.7 (4.4) | 4.4 (3.8) | 4.8 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change From Baseline
Description: Percent weight change form baseline; negative values indicate weight loss.
Time Frame: Baseline, 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: percentage of weight
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 63 | 68 | 70
percentage of weight
  Six months | -1.1 (3.7) | -5.6 (4.9) | -4.6 (5.8)
  Twelve months | -2.0 (4.1) | -4.5 (6.1) | -4.8 (6.1)
  Twenty-four months | -3.1 (5.2) | -4.4 (5.9) | -4.0 (5.8)
  Thirty-six months | -5.8 (7.1) | -4.4 (5.4) | -5.3 (6.4)

2. Secondary Outcome: Hemoglobin A1c: Change From Baseline
Description: Change in percentage of glycated hemoglobin. Negative values indicate HbA1c reduction (improvement) from baseline.
Time Frame: 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: units of HbA1c (%)
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 65 | 68 | 70
units of HbA1c (%)
  Six months | -0.3 (1.1) | -0.6 (0.8) | -0.5 (1.2)
  Twelve months | -0.4 (1.2) | -0.4 (0.8) | -0.2 (1.3)
  Twenty-four months | -0.2 (1.4) | -0.3 (1.3) | 0.1 (1.4)

3. Secondary Outcome: Systolic Blood Pressure: Change From Baseline
Description: Blood pressure is reported as change in systolic blood pressure only. Negative values indicate improvement.
Time Frame: 6, 12, 24, months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 66 | 68 | 70
mmHg
  Six months | 0 (14.7) | -4.0 (15) | -2.3 (14)
  Twelve months | 1.8 (16) | -1.8 (16) | -1.0 (15)
  Twenty-four months | -0.6 (16) | -3.5 (15) | -3.3 (15)

4. Secondary Outcome: Triglyceride Levels: Change From Baseline
Description: Triglycerides are measured in mg/dl. Negative values indicate improved triglyceride levels compared to baseline.
Time Frame: 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 61 | 66 | 70
mg/dl
  Six months | 12.5 (80) | -56.0 (253) | -21.3 (81)
  Twelve months | 7.9 (76) | -57.4 (259) | -1.1 (114)
  Twenty-four months | -8.6 (71) | -31.8 (228) | -4.1 (86)

5. Secondary Outcome: Diet Self-efficacy: Change From Baseline
Description: Diet Self-Efficacy Scale is scored 1-5 with higher scores denoting greater self confidence in managing diet and positive values denoting improved self-confidence in managing diet. Hickey ML, Owen SV, Froman RD. Instrument development: cardiac diet and exercise self-efficacy. Nursing research. 1992;41(6):347-351
Time Frame: 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 51 | 61 | 58
score on a scale
  Six months | -0.2 (0.7) | 0.3 (0.7) | 0.1 (0.6)
  Twelve months | -0.3 (0.8) | 0.2 (0.8) | -0.1 (0.8)
  Twenty-four months | -0.2 (0.8) | 0.3 (0.7) | -0.1 (0.8)
  Thirty-six months | -0.1 (0.9) | -0.1 (0.9) | -0.4 (0.8)

6. Secondary Outcome: Fat-related Diet Behavior: Change From Baseline.
Description: Fat-related diet behavior was scored on a scale of 1 to 5, in which lower scores indicate lower fat dietary habits. Negative values indicate a shift to lower-fat diet behavior.
  Kristal AR, Shattuck AL, Henry HJ. Patterns of dietary behavior associated with selecting diets low in fat: reliability and validity of a behavioral approach to dietary assessment. J Am Diet Assoc. 1990;90(2):214-220.
  Glasgow RE, Perry JD, Toobert DJ, Hollis JF. Brief assessments of dietary behavior in field settings. Addictive behaviors. 1996;21(2):239-247
Time Frame: Baseline, 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 53 | 62 | 59
score on a scale
  Six months | -0.1 (0.4) | -0.4 (0.5) | -0.3 (0.5)
  Twelve months | -0.2 (0.4) | -0.4 (0.5) | -0.3 (0.5)
  Twenty-four months | -0.2 (0.4) | -0.4 (0.4) | -0.4 (0.5)
  Thirty-six months | -0.3 (0.5) | -0.3 (0.4) | -0.3 (0.4)

7. Secondary Outcome: Dietary Restraint: Change From Baseline
Description: Dietary restraint was measured by the Dutch Eating Behavior Questionnaire with higher scores (1-5) denoting greater self-regulation of dietary behaviors and positive values denoting improved dietary restraint. Van Strien T, Frijters JER, Defares PB. The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International Journal of Eating Disorders. 1986;5(2):295-315.
Time Frame: Baseline, 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 54 | 62 | 59
score on a scale
  Six months | 0.4 (0.7) | 0.6 (0.6) | 0.6 (0.7)
  Twelve months | 0.5 (0.7) | 0.5 (0.6) | 0.5 (0.7)
  Twenty-four months | 0.3 (0.7) | 0.7 (0.7) | 0.6 (0.6)
  Thirty six months | 0.4 (0.4) | 0.7 (0.7) | 0.4 (0.8)

8. Secondary Outcome: Diabetes Distress: Change From Baseline
Description: Diabetes distress was measured with the Problem Areas in Diabetes Scale. The scale ranges from 0 to 100, in which higher scores indicate greater emotional distress, with a score of 40 marking the threshold for severe emotional distress. Negative values indicate reduction in diabetes-related distress.
  Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997;20(5):760-766
Time Frame: Baseline, 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 54 | 62 | 59
score on a scale
  Six months | -7.0 (17.6) | -12.4 (20.3) | -14.1 (19.4)
  Twelve months | -5.8 (18) | -14.4 (15) | -15.1 (21.9)
  Twenty-four months | -9.2 (22.8) | -13.0 (15.3) | -16.3 (20)
  Thirty-six months | -13.4 (22.9) | -14.1 (17.8) | -14.3 (18.6)

9. Secondary Outcome: Depression Score: Change From Baseline.
Description: The PHQ-8 measures depressed mood, with higher scores representing a higher degree of depressed mood and negative values indicating improvement. The range of scores is 0 to 24. Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009;114(1-3):163-173.
Time Frame: Baseline, 6, 12, 24, and 36 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 53 | 62 | 57
score on a scale
  Six months | -0.6 (4.5) | -1.0 (3.3) | -0.7 (3.1)
  Twelve months | -0.9 (4.1) | -1.2 (2.8) | -0.4 (3.7)
  Twenty-four months | -1.0 (4.3) | -0.8 (3.2) | -0.1 (3.1)
  Thirty-six months | -0.9 (5.2) | -0.7 (3.7) | 0.2 (4.3)

10. Other Pre Specified Outcome: Health Economics
Description: Total cost of intervention at 12 months taking into account intervention cost and savings from medication dose reduction. Incremental cost effectiveness and probabilistic sensitivity analyses and further details are reported in: Delahanty LM, Levy DE, Chang Y, Porneala BC, Goldman V, McCarthy J, Bissett L, Rodriguez AR, Chase B, LaRocca R, Wheeler A, Wexler DJ. Effectiveness of Lifestyle Intervention for Type 2 Diabetes in Primary Care: the REAL HEALTH-Diabetes Randomized Clinical Trial. J Gen Intern Med. 2020 Sep;35(9):2637-2646. doi: 10.1007/s11606-019-05629-9. Epub 2020 Jan 21. PMID: 31965526; PMCID: PMC7458982.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: US Dollar
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
Number analyzed (Participants) | 64 | 69 | 70
US Dollar | 591 [162 to 1005] | 1390 [962 to 1772] | 1814 [1384 to 2266]

ADVERSE EVENTS:
Time Frame: 3 years
Description: SAEs were collected according to standard definitions (hospitalized events, death, etc). Other Adverse events were not monitored/addressed in this lifestyle intervention study.
Arm/Group | Medical Nutrition Therapy (MNT) | In Person Group (IP) | Telephone Conference Call Group (TCC)
All-Cause Mortality (participants affected / at risk) | 1/66 | 0/70 | 1/72
Serious Adverse Events (participants affected / at risk) | 18/66 | 16/70 | 12/72
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Nutrition Therapy (MNT) (N=66) | In Person Group (IP) (N=70) | Telephone Conference Call Group (TCC) (N=72)
Hospital admission (General disorders) | 18 (25) | 16 (17) | 12 (16) — For this lifestyle intervention study, we tracked al hospital admissions as SAEs. None of the SAEs were deemed to be related to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT02320253/Prot_SAP_000.pdf